CLINICAL TRIAL: NCT02535260
Title: Clearblue Advanced Fertility Monitor Consumer Three Cycle at Home Study
Status: Withdrawn | Type: Observational
Why Stopped: Study not started, no longer required
Sponsor: SPD Development Company Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: PROTOCOL-0682
Record Dates: First submitted 2013-09-18; First posted 2015-08-28 (Estimated); Last update posted 2019-02-08 (Actual); Status verified 2019-02

CONDITIONS: Pregnancy
Keywords: Pregnancy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine samples collected throughout study
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Fertility Monitor: Clearblue Fertility Monitor

SUMMARY:
This study will assess the use of the new Clearblue Advanced Fertility Monitor in a home setting for three menstrual cycles or until pregnancy is achieved (whichever comes first) by female volunteers seeking to get pregnant.

DETAILED DESCRIPTION:
The Clearblue Fertility Monitor is a personal monitor designed to be used with disposable test sticks for the semi-quantitative measurement of estrone-3-glucuronide (E3G) and luteinising hormone (LH) in women's urine. This personal information allows women to identify their fertile window and appropriately time intercourse in order to maximise their chances of conception. A new version of this monitor (Clearblue Advance Fertility Monitor) has been developed with enhanced functionality including the option to test for pregnancy.

This study will assess the use of the new Clearblue Advanced Fertility Monitor in a home setting by female volunteers seeking to become pregnant, for three menstrual cycles or until pregnancy is achieved (whichever comes first). This is a single centre clinical study which will be conducted by volunteers at their residence and co-ordinated by the clinical department at SPD Development Company Ltd.

The overall objective of the study will be to demonstrate the usage of the new Clearblue Advanced Fertility Monitor in a home setting, to assess the benefits of monitor usage and to compare monitor data to laboratory analyses on the same urine samples.

In order to achieve these objectives, a minimum of 200 female volunteers representing the target consumer will be recruited to use the new Clearblue Advanced Fertility Monitor at home as per the instructions for use. This will involve them setting up the monitor, using the monitor for the duration of the study..

All volunteers will be required to complete a daily diary and to collect a daily urine sample. Volunteers who become pregnant on the study will be asked to continue to collect urine samples. At the end of the study all volunteers will complete a study questionnaire which includes questions relating to monitor usage and knowledge and behaviour regarding conception. Upon return to SPD, the urine samples will be tested by auto-analyser for various hormones.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Aged 18 - 45 years
* Willing to provide written informed consent to participate in the study and comply to the investigational procedures
* Naive to similar marketed products including current Clearblue Fertility Monitor and Persona
* Two natural cycles immediately prior to entering the study, each lasting between 21 and 42 days
* Seeking to become pregnant

Exclusion Criteria:

* Employees of SPD, Proctor & Gamble or Alere
* Have a condition that is known to be contra-indicated in pregnancy
* Usually have menstrual cycles which are shorter than 21 days or longer than 42 days
* Trying to conceive for12 months (for volunteers under 35) or trying to conceive for >6 months ( for volunteers 35 or older)
* Using or have used in their last 2 cycles, hormonal contraceptives including oral, emergency oral, implants, patches, transdermal injections, vaginal ring and progesterone intrauterine systems (IUS)
* Using or have used in the last 2 cycles, infertility medications or hormone replacement therapy containing hCG or LH
* Taking clomiphene citrate or other ovulation induction drugs
* Using any treatment which may affect the menstrual cycle
* Have recently been pregnant, miscarried or breastfeeding
* Have been diagnosed with polycystic ovarian syndrome (PCOS)
* Are peri- or post-menopausal e.g. experiencing symptoms such as irregular menstrual periods, hot flushes, night sweats, sleep disturbances and mood swings
* Are taking antibiotics containing tetracyclines
* Have impaired liver or kidney function
* Have previously participated in a SPD 'trying to conceive' study

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: women wishing to become pregnant
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Primary Completion 2014-04-11 (Actual)

PRIMARY OUTCOMES:
Behavioural change | 3 months
  To compare change in behaviour from self-reported baseline behaviour to that reported in daily diaries including intercourse frequency, personal fertility knowledge and pregnancy testing behaviour
Behavioural change | 3 months
  To observe % compliance of conducting tests
User comprehension | 3 months
  To assess user comprehension of the Instructions for use
Product performance | 3 months
  To assess performance of the Clearblue Advanced Fertility Monitor at identification of fertile window in relation to quantitative LH and E3G measurements
product performance | 3 months
  To compare pregnancy test results to quantitative hCG concentration

SECONDARY OUTCOMES:
Behavioural change | 3 month
  To examine pregnancy test results qualitative assessment of women's behaviour in monitor usage following early pregnancy loss, should this occur during the study
Pregnancy rate | 3 months
  To examine pregnancy rate in relation to baseline demographics, intercourse pattern during the study and expected pregnancy rate based on published literature

CONTACTS AND LOCATIONS:
Locations (1):
- SPD Development Company Ltd, Bedford, Bedfordshire, United Kingdom